CLINICAL TRIAL: NCT01761942
Title: A 10-week Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Omega-3 Fatty Acids Oral Capsules Compared With Placebo in the Treatment of Anorexia Nervosa
Brief Title: Fatty Acids Omega -3 Diet Supplementation Efficiency and Safety Evaluation in Anorexia Nervosa
Acronym: FASAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Principal Investigator, Agnieszka Piróg-Balcerzak, MD, psychiatrist, Institute of Psychiatry and Neurology, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/2011; 22/2011 (Other: Institute of Psychiatry and Neurology Warsaw)
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Anorexia Nervosa
Keywords: omega-3 fatty acids; anorexia nervosa; efficacy; safety
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo ,anorexia nervosa (Placebo Comparator): 2x3 placebo capsules with olive oil
- fatty acids preparation- eye-q (Experimental): 2 x 3 tablets of eye -q preparation daily ( 558 mg of EPA, 175 mg of DHA, 60 mg fo GLA).
  Interventions: Dietary Supplement: fatty acids preparation- eye-q

INTERVENTIONS:
Dietary Supplement: fatty acids preparation- eye-q — 3x2 tablets daily by 70 days
  Arms: fatty acids preparation- eye-q

SUMMARY:
The purpose of this study is to determine whether omega -3 fatty acids are effective and safe in treating anorexia nervosa.

DETAILED DESCRIPTION:
10-week, randomized, placebo-controlled, parallel-group study to compare the efficacy and safety of omega-3 fatty acids with placebo in the treatment of anorexia nervosa. Patients will be randomly assigned to blinded study treatment. Double-blind treatment will be preceded by a medication washout period of 1-28 days if necessary. Some patients may be taking anti-depressants or anti-psychotics, e.g. fluoxetine, prior to admission to the study. In such case the wash out period will depend on the medical treatment (dependent on the drug given) given prior to qualification to the study. Patient will be treated as inpatients during 10 weeks of the study. The study will recruit female inpatients with anorexia nervosa (aged 12 to 19 years), with DSM-IV and ICD-10 diagnosis of anorexia nervosa.BMI below 5 percentile and EAT-26 score > 30 is required at both screening and randomization.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa (DSM IV,ICD-10)
* Female
* Age 12-19
* Written informed consent given by patient and his parents

Exclusion Criteria:

* Lack of informed consent

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Omega-3 fatty acids are superior to placebo in increasing BMI at day 70 compared with baseline | day 70th
  The primary objective of this study is to compare the efficacy of EPA fatty acids with that of placebo as add-on treatment for inpatients with anorexia nervosa, as assessed by the change from baseline to day 70 in BMI (body mass index)

SECONDARY OUTCOMES:
reducing EAT -26 | day 70th
  1. To compare the effects of omega-3/6 fatty acids with the effect of placebo in reducing EAT-26 (Eating Attitude Test-26) total score at day 70 compared with baseline
changes in CGI | day 70th
  to compare the effects of fatty acids with the effect of placebo by change from baseline to day 70 in CGI (Clinical Global Impression)
change in HDRS | day 70 th
  to compare the effects of fatty acids with the effect of placebo on change form baseline to day 70 in Hamilton Depression Rating Scale
changes in BDI | day 70th
  to compare the effects of fatty acids with the effect of placebo by change form baseline to day 70 in Beck Depression Inventory
changes in YBOCS | day 70 th
  to compare the effects of fatty acids with the effect of placebo by changes in Yale-Brown Obsessive-Compulsive Scale
changes in YBOCS | day 70th
  to compare the effects of fatty acids with the effect of placebo by change form baseline to day 70 Yale-Brown Obsessive-Compulsive Scale
adverse events | 70 days time
  to evaluate the safety and tolerability of omega-3 fatty acids compared with placebo in the treatment of anorexia nervosa, as assessed by incidence and nature of adverse events
clinical laboratory tests | day 70 th
  to evaluate the safety and tolerability of omega-3 fatty acids compared with placebo in the treatment of anorexia nervosa, as assessed by changes from baseline to day 70 in clinical laboratory tests (lipids metabolism - triglycerides, HDL and LDL cholesterol)

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Piróg-Balcerzak, MD, Principal Investigator — Institute of Psychiatry and Neurology, Warsaw
Locations (1):
- Institute of Psychiatry and Neurology,, Warsaw, Masovian Voivodeship, Poland